CLINICAL TRIAL: NCT02218814
Title: Prospective, Double-blind, Randomized Study to Evaluate a Single Shot Adductor Canal Nerve Block Versus Femoral Nerve Block Combined With LIA (Local Infiltration Analgesia): Early Postoperative Period Functional Outcomes After Total Knee Replacement
Brief Title: Study to Evaluate ACB Versus FNB Early Postoperative Period Functional Outcomes After TKA
Acronym: ACB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Macrinici (Other)
Collaborators: Associated Anesthesiologists of Joliet (Unknown); Statking Consulting, Inc. (Industry)
Responsible Party: Sponsor-Investigator, George Macrinici, Physician, Presence Saint Joseph Medical Center
Organization: Presence Saint Joseph Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10231969
Record Dates: First submitted 2014-08-01; First posted 2014-08-18 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Arthroplasty, Replacement, Knee; Nerve Block
Keywords: Femoral Nerve Block; Adductor Canal Nerve Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor Canal Block: (Experimental): Adductor Canal Nerve Block: The patient is placed in a supine position with the extremity to be blocked slightly externally rotated. On the medial thigh, at the midpoint between the inguinal crease and the medial condyle, 13-6-MHz linear ultrasound transducer (SonoSite HFL38x; Washington, US) is placed in a transverse orientation to visualize the femoral artery in short axis deep to the sartorius muscle. Sterile field and patient sedation achieved. A 21-gauge,100 mm, short-bevel needle (Stimuplex; B Braun) is inserted under ultrasound guidance in in-plane technique to position the needle tip anterolateral to the artery and just deep to the posterior fascia of the sartorius muscle. Once in position, 30 mL of Bupivacaine (100 mg) is deposited adjacent to the femoral artery and deep to the Sartorius muscle, using intermittent aspiration. After completion of the procedure, a sterile dressing is placed over the needle insertion site.
  Interventions: Procedure: Adductor Canal Block, Bupivacaine
- Femoral Nerve Block (Active Comparator): Femoral Nerve Block. The procedure is conducted with the patient in a supine position with a 13-6 MHz linear ultrasound transducer (SonoSite HFL38x; Washington, US) applied to the skin at the level of the inguinal crease. The femoral artery, fascia iliac, and femoral nerve are visualized. Sterile field and patient sedation achieved. A 22-gauge, 50-mm, short-bevel stimulating needle (Stimuplex; B Braun, Bethlehem, Pennsylvania) connected to twitch monitor B/Braun Stimuplex DIG RC is inserted under ultrasound guidance using an in-plane technique from lateral to medial until a quadriceps motor response is elicited at a current between 0.5 and 0.2 mA with a pulse width of 0.1millisecond from a twitch monitor . After negative aspiration, 30 mL of Bupivacaine (100 mg) is deposited adjacent to the femoral nerve and deep to the fascia iliac, with intermittent aspiration. After completion of the procedure, a sterile dressing is placed over the needle insertion site.
  Interventions: Procedure: Femoral Nerve Block, Bupivacaine

INTERVENTIONS:
Procedure: Adductor Canal Block, Bupivacaine — Adductor Canal Nerve Block: Under US guidance and sterile technique 30 mL (100 mg) of Bupivacaine is deposited adjacent to the femoral artery and deep to the Sartorius muscle, using intermittent aspiration.
  Femoral Nerve Block: Under US guidance, using a twitch monitor and sterile technique, 30 ml of PF Normal Saline is deposited adjacent to the femoral artery at the level of inguinal crease.
  Other Names: ACB; Bupivacaine; FNB; Preservative Free Normal Saline
  Arms: Adductor Canal Block:
Procedure: Femoral Nerve Block, Bupivacaine — Femoral Nerve Block: Under US guidance, using a twitch monitor and sterile technique, 30 ml (100 mg) of Bupivacaine is deposited adjacent to the femoral artery at the level of inguinal crease.
  Adductor Canal Nerve Block: Under US guidance and sterile technique 30 mL of PF Normal Saline is deposited adjacent to the femoral artery and deep to the Sartorius muscle, using intermittent aspiration.
  Other Names: FNB; Bupivacaine; ACB; Preservative Free Normal Saline
  Arms: Femoral Nerve Block

SUMMARY:
The purpose of this study is to determine if patients undergoing a Total Knee Arthroplasty who receive a single shot Adductor Canal nerve block and local infiltration will have improved functional outcomes compared to individuals who receive a femoral nerve block and local infiltration during the first 24 hours post surgery.

DETAILED DESCRIPTION:
Title: Prospective, Double-blind, Randomized Study to Evaluate a Single Shot Adductor Canal Nerve Block versus Femoral Nerve Block combined with LIA (Local Infiltration Analgesia): Early Postoperative Period Functional Outcomes after Total Knee Arthroplasty.

Objectives:

Primary: To determine if patients undergoing a Total Knee Arthroplasty who receive an Adductor Canal block will result in increased quadriceps muscle strength (MVIC) compared to those who receive a Femoral Nerve block at 24 hours.

Secondary: The secondary objective is to determine whether Adductor Canal nerve block results in improved functional outcomes as evidenced by Time up and GO, Range of Motion and Six-Minute Walk Test at 24 hours, 48 hours and 6 months.

To assess post-operative pain as measured by the Visual Analog pain score (VAS) immediately prior to the start of, during, and after each in-patient physical therapy session.

Study Design: Prospective, double-blind, randomized study

Description of Intervention: The devices to be used in this study are intended for nerve blocks and consist of 13-6 MHz linear ultrasound transducer (SonoSite HFL38x; Washington, US), a 22-gauge, 50-mm, short-bevel stimulating needle (Stimuplex; B Braun, Bethlehem, Pennsylvania), B/Braun Stimuplex DIG RC, Bupivacaine HCl 100 mg injected in the Adductor Canal or around the Femoral nerve.

Femoral nerve block in combination with local infiltration analgesia is the standard of care in the investigators institution at present.

Bupivacaine HCl 100 mg in combination with Toradol 30 mg are used for local infiltration of the anterior lateral and lateral posterior side of the knee, done by the surgeon using a standard technique.

Subject Population:The study will include both male and female adults who will meet the inclusion criteria and none of exclusion criteria. For each patient time to conduct the blocks will vary between 5-10 minutes, local infiltration analgesia between 5-10 minutes, physical therapy tests between 30 minutes and one hour each encounter, VAS pain assessment between 2-5 minutes

Subject Participation Duration:The rate of patient accrual, and the prescribed follow-up time, the total duration of this study is expected to be approximately 18 months where enrollment is expected to occur over 12 months with a follow-up period of 6 months in the physical therapy office visits.

Number of Patients:The study will include 120 patients.

Number of Sites: The study will include one site.

Study Duration:The expected study duration is approximately 18 months.

Endpoints: Endpoints of this study will include quadriceps muscle strength, ROM of the knee, TUG, 6 minute walk test, knee pain score (VAS), activities of daily living, adverse events and will be studied from the baseline up to 6 month after TKR. VAS pain score will be assessed at each physical therapy encounter.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 40-80 years of age and skeletally mature
* Subject BMI is < 40
* Subject has been selected by the surgeon for TKA.
* Subject is taking less than 30 mg of Morphine per day.
* Subject is willing and able to sign a written consent form
* The subject has the mental capacity and the willingness to comply with the specified follow-up evaluations, and can be contacted by telephone by the site personnel.
* The subject is not pregnant, does not intend to become pregnant and has a significant other mirroring her intentions.

Exclusion Criteria:

* Subject is not neurologically intact (sensory, motor, and reflex deficit)
* Subject has pain in the limb scheduled for surgery that is out of proportion of expected pain usual for this pathology
* Subject scheduled for simultaneous bilateral knee replacement
* Subject has a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years
* Subject with prior reconstructive knee surgery on the operated limb
* Subject with primary bone tumor in the knee area
* Subject anticipates having a lower extremity surgery other than the investigational surgery during the course of the study
* Subject has a history of substance abuse
* Subject is currently involved in another study or have received investigational product or treatment within the last 30 days
* Subject is pregnant or planning on becoming pregnant during the study period
* Subject is accepting workers' compensation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength (MVIC) difference between the ACB and FNB after total knee arthroplasty. | Baseline, 6, 24, 48 hours and at 6 month after nerve block performance
  Maximum Voluntary Isovolumetric Contraction (MVIC) measured in Newtons of the quadriceps muscle normalized to body mass index (N•m/kg). The 6 hours post procedure percent of baseline is considered the primary clinical success criterion variable of this study.

SECONDARY OUTCOMES:
Knee range of motion | Baseline, 6, 24 48 hours and 6 month after the nerve block performance
  Knee range of motion is measured as a combined flexion/extension either actively or passively with assistance. Knee range of motion is typically measured in the supine position. The examiner will measure knee flexion passively using a goniometer. It has been validated as an outcome measure in total knee arthroplasty. To be able to navigate stairs 90 degrees of flexion is required. To adequately perform activities of daily living (ADL's), 110 degrees of flexion is required. The minimum detectable change in knee flexion for an individual is 9.6 degrees.
Time Up and Go | Baseline, 24, 48 hours and 6 month after the nerve block performance
  The TUG test records the time taken to stand up from a standard height arm chair, walk 3m, walk back to the chair, and sit down. It is meant to assess a patients balance and risk of falling. Assistive devices, for example, a walker, are allowed to be used if needed. This test has been validated as an early functional outcome after TKA. Maximum improvement occurs between the sixth and ninth postoperative weeks, with a plateau at 10 weeks. Freely independent patients are able to complete the task in 10 seconds, whereas a time greater than 30 seconds corresponds to patients being dependent in most activities. The minimum detectable change is 2.5 seconds.
6 Minute Walk Test | Baseline and at 6 month after the surgery
  The 6-Minute Walk Test (6MWT) records the maximum distance ambulated on level ground without physical assistance in six minutes with standardized encouragement. It has been validated for evaluation of functional outcome after TKA. Assistive devices are allowed if needed. The minimum distance that is required to perform ADL's is 300m. After TKA, increase in 6MWT distance typically follow pattern where maximal improvement occurs in the first 12 weeks postoperatively, specifically between weeks 6 and 9, followed by a slower improvement between weeks 12 and 26, reaching a plateau at 26 weeks. The minimum detectable change (MDC) for the 6MWT is reported to be 61.3m.

CONTACTS AND LOCATIONS:
Overall Officials: George I Macrinici, MD, Principal Investigator — Presence Saint Joseph Medical Center
Locations (1):
- Presence Saint Joseph Medical Center, Joliet, Illinois, United States

REFERENCES:
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Chaumeron A, Audy D, Drolet P, Lavigne M, Vendittoli PA. Periarticular injection in knee arthroplasty improves quadriceps function. Clin Orthop Relat Res. 2013 Jul;471(7):2284-95. doi: 10.1007/s11999-013-2928-4. Epub 2013 Mar 21. PMID 23516031
- [Background] Wasserstein D, Farlinger C, Brull R, Mahomed N, Gandhi R. Advanced age, obesity and continuous femoral nerve blockade are independent risk factors for inpatient falls after primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1121-4. doi: 10.1016/j.arth.2012.08.018. Epub 2012 Dec 21. PMID 23265274
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Andersen HL, Gyrn J, Moller L, Christensen B, Zaric D. Continuous saphenous nerve block as supplement to single-dose local infiltration analgesia for postoperative pain management after total knee arthroplasty. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):106-11. doi: 10.1097/AAP.0b013e31827900a9. PMID 23222363
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Andersen LO, Gaarn-Larsen L, Kristensen BB, Husted H, Otte KS, Kehlet H. Analgesic efficacy of local anaesthetic wound administration in knee arthroplasty: volume vs concentration. Anaesthesia. 2010 Oct;65(10):984-90. doi: 10.1111/j.1365-2044.2010.06452.x. PMID 20649528
- [Background] Andersen LO, Husted H, Kristensen BB, Otte KS, Gaarn-Larsen L, Kehlet H. Analgesic efficacy of subcutaneous local anaesthetic wound infiltration in bilateral knee arthroplasty: a randomised, placebo-controlled, double-blind trial. Acta Anaesthesiol Scand. 2010 May;54(5):543-8. doi: 10.1111/j.1399-6576.2009.02196.x. Epub 2010 Jan 6. PMID 20055763
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738
- [Derived] Macrinici GI, Murphy C, Christman L, Drescher M, Hughes B, Macrinici V, Diab G. Prospective, Double-Blind, Randomized Study to Evaluate Single-Injection Adductor Canal Nerve Block Versus Femoral Nerve Block: Postoperative Functional Outcomes After Total Knee Arthroplasty. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):10-16. doi: 10.1097/AAP.0000000000000507. PMID 27811526
- See also: Bupivacaine — http://www.accessdata.fda.gov/drugsatfda_docs/label/2012/018692s015lbl.pdf